CLINICAL TRIAL: NCT03117361
Title: Phase II Trial of Plitidepsin (Aplidin®) in Combination With Bortezomib and Dexamethasone in Multiple Myeloma Patients Double Refractory to Bortezomib and Lenalidomide
Brief Title: Trial of Plitidepsin (Aplidin®) in Combination With Bortezomib and Dexamethasone in Multiple Myeloma Patients Double Refractory to Bortezomib and Lenalidomide
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PharmaMar has decided to end this study due to the slow recruitment rate of the trial
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-B-022-15
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; plitidepsin; Aplidin
MeSH Terms: conditions — Multiple Myeloma | interventions — plitidepsin; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Plitidepsin + bortezomib + dexamethasone
  Plitidepsin will be administered as a 3-hour intravenous (i.v.) infusion on Day(D) 1 and 15 , every four weeks (q4wk)
  Bortezomib will be administered as a bolus subcutaneous (s.c.) injection on D 1, 4, 8 and 11,q4wk
  Dexamethasone will be taken orally on D1,8,15 and 22, q4wk
  Interventions: Drug: plitidepsin; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: plitidepsin — Patients received plitidepsin as a 3-hour i.v. infusion at a dose of 5 mg/m2 on Days 1 and 15 every Four Weeks.
Drug: Bortezomib — BTZ as a 3-5 second bolus s.c. injection at a dose of 1.3 mg/m2 on Days 1, 4, 8 and 11 every four weeks
Drug: Dexamethasone — DXM orally at a dose of 40 mg/day on Days 1, 8, 15 and 22 every four weeks

SUMMARY:
This is a multi-center, open-label, single arm, non-comparative phase II trial, designed to evaluate the efficacy of plitidepsin in combination with bortezomib and dexamethasone in patients with Multiple Myeloma (MM) double refractory to bortezomib and lenalidomide.

DETAILED DESCRIPTION:
This is a multi-center, open-label, single arm, non-comparative phase II trial, designed to evaluate the efficacy of plitidepsin in combination with bortezomib and dexamethasone in patients with MM double refractory to bortezomib and lenalidomide.The primary endpoint will be overall response rate (ORR), including stringent complete response (sCR), complete response (CR), very good partial response (VGPR) and partial response (PR).

Approximately 64 evaluable patients will be needed for the evaluation of the primary endpoint, ORR.

An early futility analysis will be performed with the efficacy data collected from the first 20 evaluable patients. The futility analysis will commence once patient number 20 has completed two full treatment cycles. Patient recruitment will not be halted during the conduct of this futility analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written informed consent (IC) in accordance with institutional and local guidelines.
2. Age ≥ 18 years.
3. Patients must have a confirmed diagnosis of MM according to the Durie and Salmon criteria.
4. Patients must have measurable disease defined as any of the following:

   1. Serum M-protein ≥ 0.5 g/dL or ≥ 0.2 g/24-h urine light chain (UFLC) excretion.
   2. In patients who lack measureable M-protein in serum or urine, i.e., serum M-protein < 0.5 g/dL and urine M-protein < 0.2 g/24 h, serum free light chain (SFLC) levels are most informative. SFLC levels can be used only if the baseline SFLC ratio is abnormal (<0.26 or >1.65), indicating clonality. In addition, the baseline SFLC level must be ≥10 mg/dl of the appropriate involved light chain isotype.
   3. When applicable, measurable soft tissue plasmacytoma ≥ 2 cm, by either physical examination and/or applicable radiological evaluation (i.e., magnetic resonance imaging [MRI], computed tomography [CT]-scan).
5. Prior autologous and/or allogeneic hematopoietic stem cell transplantation (HSCT) patients are allowed. Patients must not have acute/chronic graft-versus-host disease (GVHD) or be receiving immunosuppressive therapy at least 90 days before the onset of treatment with the trial drug(s).
6. Patients must have received previous treatment with bortezomib and lenalidomide and be refractory to both.
7. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
8. Recovery to grade ≤ 1 from any non-hematological adverse event (AE) derived from previous treatment (if present, alopecia and peripheral neuropathy must be grade <1).
9. Laboratory data:

   1. Hemoglobin ≥ 8 g/dL.
   2. Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3 (1.0 x 109/L) (≥ 0.5 x 109/L if due to extensive bone marrow [BM] involvement by ≥ 50% of plasma cells in BM biopsy). Screening of ANC should be independent of granulocyte- and granulocyte/macrophage-colony stimulating factor (G-CSF and GM-CSF) support for at least one week and of pegylated G-CSF for at least two weeks.
   3. Platelet count ≥ 50,000/mm3 (50.0 x 109/L) for patients in whom < 50% of the BM nucleated cells are plasma cells.
   4. Platelet count ≥ 25,000/mm3 (25.0 x 109/L) for patients in whom ≥ 50% of BM nucleated cells are plasma cells.
   5. Serum total bilirubin < 1.5 x institutional upper limit of normal (ULN) (except when Gilbert syndrome is clearly documented and other liver function tests are within normal levels).
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x institutional ULN and alkaline phosphatase (AP) ≤ 2.5 x institutional ULN.
   7. Creatinine clearance (CrCl) > 30 mL/min, measured or calculated according to Cockcroft and Gault's formula.
   8. Albumin ≥ 2.5 g/dl.
10. Evidence of non-childbearing status for women of childbearing potential (WOCBP): WOCBP must have a negative serum or urine pregnancy test within seven days prior to enrolment and must agree to use a highly effective contraceptive measure throughout the trial and during six months after treatment discontinuation. Male patients enrolled in the study should also use contraceptive methods during and after treatment discontinuation.
11. Left ventricular ejection fraction (LVEF) ≥ 45%.
12. Patients must have a BM assessment within three weeks prior to enrolment.

Exclusion Criteria:

1. Previous treatment with plitidepsin.
2. Active or metastatic primary malignancy other than MM.
3. Serious concomitant systemic disorders that would compromise the safety of the patient or the patient's ability to complete the trial, including the following specific conditions:

   1. Uncontrolled psychiatric illness or medical illness that the Investigator feels will compromise the patient's tolerance of the trial medication.
   2. Significant non-neoplastic liver disease.
   3. Uncontrolled endocrine diseases (i.e., requiring relevant changes in medication within the last month, or hospital admission within the last three months).
   4. Uncontrolled systemic infection.
   5. Acute infiltrative pulmonary and pericardial disease.
4. Other relevant cardiac conditions:

   1. Symptomatic arrhythmia (excluding anemia-related grade ≤ 2 sinusal tachycardia) or any arrhythmia requiring ongoing treatment, and/or prolonged grade ≥ 2 QT-QTc; or presence of unstable atrial fibrillation (according to the National Cancer Institute Common Terminology Criteria for the Classification of Adverse Events [NCI-CTCAE] v4.0). Patients on treatment for stable atrial fibrillation are allowed, provided they do not meet any other cardiac or prohibited drug exclusion criterion.
   2. History or presence of unstable angina, myocardial infarction, valvular heart disease, cardiac amyloidosis or congestive heart failure within the last 12 months.
   3. Uncontrolled arterial hypertension (≥ 150/100 mmHg) despite optimal medical therapy.
   4. Previous treatment with doxorubicin at cumulative doses of > 400 mg/m², or equivalent.
5. History of hypersensitivity reactions and/or intolerance to bortezomib, polyoxyl 35 castor oil, mannitol, boron or dexamethasone.
6. Myopathy or any clinical situation that causes significant and persistent elevation of creatine phosphokinase (CPK) (> 2.5 ULN) in two different determinations performed within one week of each other.
7. Grade ≥ 1 neuropathy (either bortezomib-related or not) according to NCI-CTCAE v4.0.
8. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patients' participation in this trial.
9. Pregnant and/or lactating women.
10. Known active human immunodeficiency virus (HIV) infection (HIV testing is not required unless infection is clinically suspected).
11. Active hepatitis B or C virus (HBV or HCV) infection.
12. Treatment with any Investigational Medicinal Product (IMP) in the 30 days before inclusion in the trial.
13. Concomitant medications that include corticosteroids, chemotherapy (CT), or other therapy that is or may be active against myeloma. Concurrent corticosteroids are allowed as an equivalent to a prednisone dose of ≤ 10 mg daily, administered as an antiemetic or as premedication for blood products.
14. Wash-out periods after the end of the previous therapy:

    1. Nitrosoureas must be discontinued six weeks prior to Cycle (C) 1, D1.
    2. Thirty days for other CTs and 15 days for other biological agents prior to C1 D1.
    3. Thirty days after the end of any prior radiation or radionuclide therapy (six weeks in the case of prior extensive external beam radiation, with more than 25% of BM distribution).
15. Plasma cell leukemia at the time of trial entry.
16. Disease-related symptomatic hypercalcemia despite optimal medical therapy.
17. Limitation of the patient's ability to comply with the treatment or follow-up protocol.
18. Contraindication to use steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- France (2):
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - Institut Gustave Roussy, Villejuif
- Italy (3):
  - Policlinico Vittorio Emanuele Hospital, Catania
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Spain (8):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Institut Català d´Oncologia Girona, Girona
  - Institut Català d´Oncologia L´Hospitalet, L'Hospitalet de Llobregat
  - Hospital General Universitario J.M. Morales Meseguer, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Complejo Hospitalario Regional Virgen Del Rocio, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients participated between 15May2017 - 30Jul2018 (last follow-up cutoff date). The 1st dose/1st cycle was administered on 15May2017 and the last dose/last cycle on 23Jul2018. At cutoff date 10 patients had been included and treated with plitidepsin+BTZ+DXM and they were evaluable for safety. 8 of these were evaluable for the efficacy endpoint
Pre-assignment Details: IC signed;Age≥18 years;confirmed diagnosis of MM,ECOG PS≤2;LVEF≥45%;negative pregnancy test
Groups:
- Experimental: Plitidepsin was to be administered as a 3-hour (h) intravenous (i.v.) infusion at a dose of 5 mg/m2, on Day (D) 1 and 15, every four weeks (q4wk); BTZ was to be administered as a subcutaneous (s.c.) injection at a dose of 1.3 mg/m2 on D1, 4, 8 and 11, q4wk and DXM was to be taken orally at a dose of 40 mg/day on D1, 8, 15 and 22, q4wk. A cycle was defined as 28 days, plus any additional days required for dosing delays due to any reason. Treatment cycles were repeated q4wk.
Period: Overall Study
Arm/Group | Experimental
Started | 10
Completed | 0
Not Completed | 10
Not completed — Progressive disease | 5
Not completed — Death | 1
Not completed — Physician Decision | 2
Not completed — On study treatment at the end of study | 1
Not completed — Treatment-related adverse event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 59 [43 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7
  Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 4
  France | 3
  Spain | 3
ECOG PS [Count of Participants; unit: Participants] — ECOG PS, Eastern Cooperative Oncology Group performance status PS 0 Fully active able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities up and about more than 50% of waking hours PS 3 Capable of only limited selfcare confined to bed or chair more than 50% of waking hours PS 4 Completely disabled cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    PS 0 | 5
    PS 1 | 4
    PS 2 | 1
Multiple myeloma type at diagnosis [Count of Participants; unit: Participants]
  Secretory IgA | 2
  Secretory IgG | 4
  Secretory Kappa light-chain disease | 2
  Secretory Lambda light-chain disease | 2
Durie-Salmon stage and subclassification at diagnosis [Count of Participants; unit: Participants] — 4 patients had missing data in stage and sub-classification Stage I: All of the following: Hemoglobin>10 g/dl,Serum calcium<10.5 mg/dL, normal bone structure,IgG<5 g/dL; IgA<3 g/dL, Urine light chain M-component<4 g/24h Stage II:Fitting neither Stage I nor Stage III Stage III: One or more of the following: Hemoglobin<8.5 g/dL, Serum calcium>12 mg/dL,Advanced lytic bone lesions,IgG>7 g/dL; IgA> 5 g/dL,Urine light chain M-component>12 g/24h Subclassification: A, serum creatinine<2.0 mg/dL;B, serum creatinine>2.0 mg/dL
  Participants
    IIA | 2
    IIIA | 3
    IIIB | 1
    Missing | 4
ISS stage at diagnosis [Count of Participants; unit: Participants] — ISS, International Staging System ISS stage I was defined as serum β2-microglobulin level less than 3.5 mg/L and serum albumin level ≥ 3.5 g/dL. ISS stage II included all patients with neither stage I nor stage III disease. ISS stage III was defined as serum β2-microglobulin level ≥ 5.5 mg/L, irrespective of serum albumin level
  Participants
    ISS I | 1
    ISS II | 1
    ISS III | 4
    Not done | 4
R-ISS stage at study entry [Count of Participants; unit: Participants] — R-ISS, Revised International Staging System Stage I: Serum β2 microglobulin<3.5 mg/l; Serum albumin≥3.5 g/dl;Standard-risk chromosomal abnormalities (CA);Normal LDH Stage II: Not R-ISS stage I or III Stage III: Serum β2 microglobulin≥5.5 mg/L and either High-risk CA by FISH OR High LDH
  Participants
    Stage II | 3
    Stage III | 3
    Non available genetic results | 4
Cytogenetic at study entry [Count of Participants; unit: Participants]
  High risk | 2
  Standard risk | 4
  Non available genetic results | 4
Disease status with respect to last prior therapy [Count of Participants; unit: Participants] — Total refractory MM included 2 categories of refractory:
  * Primary Refractory: disease that was non-responsive in patients who had never achieved a MR or better, with any therapy. It included patients who never achieved MR or better, in whom there was no significant change in M-protein and no evidence of clinical progression, as well as primary, refractory PD where patients met criteria for true PD.
  * Relapsed and refractory: disease that was non-responsive while on salvage therapy, or progressed within 60 days of the last therapy in patients who had achieved MR or better at some point
  Participants
    Primary Refractory | 7
    Relapsed and refractory | 3
Best response to last prior anticancer therapy [Count of Participants; unit: Participants] — Partial response (PR): had ≥50% reduction in serum M-protein and reduction of 24-hour urine M-protein by 90% or to <200 mg/24h Minimal response (MR): had ≥25% but ≤49% reduction of serum M-protein and reduction of 24h urine M-protein 50-89%.
  Progressive disease (PD): had a 25% increase from the lowest response value in any of the following: serum M-protein, urine M-protein, BM plasma cell percentage, or difference in the kappa and lambda FLC. PD also diagnosed when an increase size or new bone lesions Stable disease (SD): not meet the criteria for PR, MR or PD
  Participants
    PR | 2
    MR | 1
    SD | 2
    PD | 5
Prior HSCT [Count of Participants; unit: Participants] — HSCT, hematopoietic stem cell transplantation
  Participants
    Autologous | 6
    Autologous and allogenic | 2
    No | 2
Lines of prior chemotherapy [Count of Participants; unit: Participants]
  3 lines | 1
  4 lines | 2
  5 lines | 4
  8 lines | 2
  9 lines | 1
Weight [Median (Full Range); unit: kg] | 71.4 [51.0 to 105.3]
Height [Median (Full Range); unit: cm] | 167.1 [152 to 186]
Body surface area [Median (Full Range); unit: m^2] | 1.8 [1.5 to 2.2]
Time from diagnosis to first plitidepsin infusion [Median (Full Range); unit: months] | 70.7 [16 to 168]
Time from last progressive disease to first infusion [Median (Full Range); unit: weeks] | 5.3 [2 to 14]
Lines of prior chemotherapy [Median (Full Range); unit: Lines] | 5 [3 to 9]
Agents of prior chemotherapy [Median (Full Range); unit: Agents] | 9 [5 to 13]
TTP to last anticancer therapy [Median (Full Range); unit: months] — Time to progression (TTP) was defined as the time, in months, from the date of the first infusion of last anticancer therapy to the date of documented PD previous study entry.
  months | 3.4 [1.6 to 10.6]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Partial response (PR): ≥50% reduction in serum M-protein and reduction of 24-hour urine M-protein by 90% or to <200 mg/24h Minimal response (MR): ≥25% but ≤49% reduction of serum M-protein and reduction of 24h urine M-protein 50-89%.
  Progressive disease (PD): 25% increase from the lowest response value in any of the following: serum M-protein, urine M-protein, BM plasma cell percentage, or difference in the kappa and lambda FLC. PD also diagnosed when an increase size or new bone lesions Stable disease (SD): not meet the criteria for PR, MR or PD Primary analysis should have been done once a total of 64 patients have received plitidepsin+BTZ+DXM with one futility analysis planned after the inclusion of 20 evaluable patients that had completed two full treatment cycles. Only 10 patients were treatedand 8 evaluable for the primary endpoint (ORR according to IMWG criteria). As a result of slow patient accrual, the study was closed before reaching the target enrollment
Time Frame: From the date of first drug administration to the date of at least one disease assessment, up to 100 weeks
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
Participants
  PR | 1
  MR | 1
  SD | 5
  PD | 1

2. Primary Outcome: Overall Response Rate
Description: The primary endpoint was overall response rate (ORR) (including stringent complete response [sCR], complete response [CR], very good partial response [VGPR] and partial response [PR]), according to the IMWG response criteria.
Time Frame: From the date of first drug administration to the date of at least one disease assessment, up to 100 weeks
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 12.5 [0.3 to 52.7]

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate defined as minimal response or better
Time Frame: From the date of first drug administration to the date of at least one disease assessment, up to 100 weeks
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 25.0 [3.2 to 65.1]

4. Secondary Outcome: Disease Control Rate
Description: Disease control rate defined as stable disease [SD] or better
Time Frame: From the date of first drug administration to the date of at least one disease assessment, up to 100 weeks
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 87.5 [47.3 to 99.7]

5. Secondary Outcome: Duration of Response
Description: Duration of Response defined as the time, in months, from the date of first documentation of response to the date of disease progression. Response was assessed according to the IMWG classification response criteria.
Time Frame: From the date of first documentation of response to the date of disease progression, up to 100 weeks
Population: Only one patient achieved a partial response
Measure: Number; unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 1
months | 9.2

6. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) was defined as the time, in months, from the date of the first infusion to the date of documented PD or death due to PD. TTP was to be censored on the date of the last tumor assessment or on the date of the first drug administration if there were no tumor assessments.
  Progressive disease (PD): 25% increase from the lowest response value in any of the following: serum M-protein, urine M-protein, BM plasma cell percentage, or difference in the kappa and lambda FLC. PD also diagnosed when an increase size or new bone lesions.
Time Frame: From the date of the first infusion to the date of documented PD or death due to PD, up to 100 weeks
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 8
months | 2.7 [0.7 to NA] — upper limit was not estimable due to few participants with events

7. Secondary Outcome: Percentage of Participants With Progression Disease at 3 Months
Description: Progression disease was defined as documented PD or death due to PD Progressive disease (PD): 25% increase from the lowest response value in any of the following: serum M-protein, urine M-protein, BM plasma cell percentage, or difference in the kappa and lambda FLC. PD also diagnosed when an increase size or new bone lesions.
Time Frame: From the date of the first infusion to the date of documented PD or death due to PD, up to 3 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 37.5 [4.0 to 71.0]

8. Secondary Outcome: Percentage of Participants With Progression Disease at 6 Months
Description: Progression disease was defined as documented PD or death due to PD. Progressive disease (PD): 25% increase from the lowest response value in any of the following: serum M-protein, urine M-protein, BM plasma cell percentage, or difference in the kappa and lambda FLC. PD also diagnosed when an increase size or new bone lesions
Time Frame: From the date of the first infusion to the date of documented PD or death due to PD, up to 6 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 25.0 [0.0 to 55.0]

9. Secondary Outcome: Percentage of Participants With Progression Disease at 12 Months
Description: as for outcome 8
Time Frame: From the date of the first infusion to the date of documented PD or death due to PD, up to 12 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 25.0 [0.0 to 55.0]

10. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time, in months, from the date of first drug administration to the date of documented PD, or death (of any cause). If any patient was lost to follow-up before PD or received another antitumor therapy, PFS was to be censored on the date of the last tumor assessment. If there were no tumor assessments, these parameters were to be censored on the date of the first drug administration.
  Progressive disease (PD): 25% increase from the lowest response value in any of the following: serum M-protein, urine M-protein, BM plasma cell percentage, or difference in the kappa and lambda FLC. PD also diagnosed when an increase size or new bone lesions.
Time Frame: From the date of first drug administration to the date of documented PD, or death (of any cause), up to 100 weeks
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 8
months | 2.7 [0.7 to NA] — upper limit was not estimable due to few participants with events

11. Secondary Outcome: Percentage of Participants With Progression-free Survival at 3 Months
Description: Progression-free Survival was defined as documented PD, or death of any cause. Progressive disease (PD): 25% increase from the lowest response value in any of the following: serum M-protein, urine M-protein, BM plasma cell percentage, or difference in the kappa and lambda FLC. PD also diagnosed when an increase size or new bone lesions.
Time Frame: From the date of first drug administration to the date of documented PD, or death (of any cause), up to 3 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 37.5 [4.0 to 71.0]

12. Secondary Outcome: Percentage of Participants With Progression-free Survival at 6 Months
Description: as for outcome 11
Time Frame: From the date of first drug administration to the date of documented PD, or death (of any cause), up to 6 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 25.0 [0.0 to 55.0]

13. Secondary Outcome: Percentage of Participants With Progression-free Survival at 12 Months
Description: Progression-free survival (PFS) was defined as the time, in months, from the date of first drug administration to the date of documented PD, or death (of any cause). If any patient was lost to follow-up before PD or received another antitumor therapy, PFS was to be censored on the date of the last tumor assessment. If there were no tumor assessments, these parameters were to be censored on the date of the first drug administration Progressive disease (PD): 25% increase from the lowest response value in any of the following: serum M-protein, urine M-protein, BM plasma cell percentage, or difference in the kappa and lambda FLC. PD also diagnosed when an increase size or new bone lesions.
Time Frame: From the date of first drug administration to the date of documented PD, or death (of any cause), up to 12 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 25.0 [0.0 to 55.0]

14. Secondary Outcome: Event-free Survival
Description: Event-free survival (EFS) was defined as the time, in months, from the date of first drug administration to the date of onset of the first drug-related event leading to treatment discontinuation, documented PD or death. The censoring rules defined above for PFS were used for EFS
Time Frame: From the date of first drug administration to the date of onset of the first drug-related event leading to treatment discontinuation, documented PD or death, up to 100 weeks
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 8
months | 2.7 [0.7 to NA] — upper limit was not estimable due to few participants with events

15. Secondary Outcome: Percentage of Participants With Event-free Survival at 3 Months
Description: Event-free survival (EFS) was defined as the first drug-related event leading to treatment discontinuation, documented PD or death.
  rogressive disease (PD): 25% increase from the lowest response value in any of the following: serum M-protein, urine M-protein, BM plasma cell percentage, or difference in the kappa and lambda FLC. PD also diagnosed when an increase size or new bone lesions.
Time Frame: From the date of first drug administration to the date of onset of the first drug-related event leading to treatment discontinuation, documented PD or death, up to 3 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 37.5 [4.0 to 71.0]

16. Secondary Outcome: Percentage of Participants With Event-free Survival at 6 Months
Description: Event-free survival (EFS) was defined as the first drug-related event leading to treatment discontinuation, documented PD or death.
  Progressive disease (PD): 25% increase from the lowest response value in any of the following: serum M-protein, urine M-protein, BM plasma cell percentage, or difference in the kappa and lambda FLC. PD also diagnosed when an increase size or new bone lesions.
Time Frame: From the date of first drug administration to the date of onset of the first drug-related event leading to treatment discontinuation, documented PD or death, up to 6 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 25.0 [0.0 to 55.0]

17. Secondary Outcome: Percentage of Participants With Event-free Survival at 12 Months
Description: as for outcome 16
Time Frame: From the date of first drug administration to the date of onset of the first drug-related event leading to treatment discontinuation, documented PD or death, up to 12 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 25.0 [0.0 to 55.0]

18. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time, in months, from the date of first drug administration to the date of death (of any cause) or last patient contact (in this case, survival was to be censored on that date).
Time Frame: From the date of first drug administration to the date of death (of any cause) or last patient contact, up to 100 weeks
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 8
months | NA [2.3 to NA] — Median and upper limit was not estimable due to few participants with events

19. Secondary Outcome: Percentage of Participants With Overall Survival at 6 Months
Description: Overall survival (OS) was defined as death of any cause.
Time Frame: From the date of first drug administration to the date of death (of any cause) or last patient contact, up to 6 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 55.6 [6.9 to 100.0]

20. Secondary Outcome: Percentage of Participants With Overall Survival at 12 Months
Description: Overall survival (OS) was defined as death of any cause.
Time Frame: From the date of first drug administration to the date of death (of any cause) or last patient contact, up to 12 months
Population: 1 died without any valid tumor assessment done
  1 discontinued treatment-related AEs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
percentage of participants | 55.6 [6.9 to 100.0]

ADVERSE EVENTS:
Time Frame: From first infusion to 30 days after the last administration of trial drug and until their resolution, an average of 2 years
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 3/10
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=10)
Haematoma (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (3)
Intramedullary rod insertion (Surgical and medical procedures) | 1 (1)
Asthenia/Fatigue (General disorders) | 4 (22)
Extravasation (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (7)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (6)
Depression (Psychiatric disorders) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (12)
Antithrombin III decreased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood cholesterol (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (3)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 6 (25)
Neutropenia (Blood and lymphatic system disorders) | 3 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (35)
Headache (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (14)
Sciatica (Nervous system disorders) | 1 (4)
Seizure (Nervous system disorders) | 1 (1)
Cataract (Eye disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (7)
Gastric disorder (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 5 (8)
Vomiting (Gastrointestinal disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (19)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Folliculitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (2)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2)

LIMITATIONS AND CAVEATS:
On 29052018 the Sponsor closed the recruitment of the study due to the slow patient accrual. Besides the negative opinion of the EMA recommending the refusal of the marketing authorization for plitidepsin for MM reinforced the decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2015-11-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT03117361/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT03117361/SAP_001.pdf